CLINICAL TRIAL: NCT02039245
Title: An Open-Label Study to Evaluate the Multiple Dose Pharmacokinetics of Canagliflozin (JNJ-28431754) and Metformin Following Once-Daily Administration of 2 Canagliflozin/Metformin XR (150/1,000-mg) Fixed Dose Combination Tablets in Healthy Subjects
Brief Title: Multiple Dose Pharmacokinetics of Canagliflozin/Metformin 150/1,000 mg Fixed Dose Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103255; 28431754DIA1042 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Canagliflozin; Metformin; INVOKANA®; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Canagliflozin/Metformin XR (Experimental): Each patient will receive 2 tablets of CANA/MET XR combination of total dose 300/2000 mg
  Interventions: Drug: CANA/MET XR FDC

INTERVENTIONS:
Drug: CANA/MET XR FDC — Each tablet contains Canagliflozin/extended release Metformin (CANA/MET XR) fixed dose combination (FDC) of 150 mg/1,000 mg, to be taken orally (by mouth)

SUMMARY:
The purpose of this study is to evaluate the multiple dose pharmacokinetics of 2 Canagliflozin/extended release Metformin (CANA/MET XR) fixed dose combination tablets (150 mg/1,000 mg each) following once-daily oral dosing in healthy participants.

DETAILED DESCRIPTION:
This is an open-label (physicians and participants know the identity of the assigned treatment), multiple-dose, single-center, pharmacokinetic study of a fixed dose combination (FDC) of 150 mg/1,000 mg Canagliflozin/extended release Metformin (CANA/MET XR) tablets. The study will consist of 3 phases: a Screening Phase of approximately 3 weeks, an Open-Label Treatment Phase, (when the participants will be confined to the study center for 11 days), and a Follow-up Phase of about 10 days. The total duration of the study will be about 42 days for each participant. During the Open-Label Treatment Phase, approximately 12 healthy adult participants will receive a single oral dose of 2 CANA/MET XR tablets once daily for 7 days after a provided dinner. Participants will be required to fast from the end of lunch until the dinner (a period of at least 6.5 hours) on Days 1 and 7 only.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document indicating they understand the purpose of the study and procedures
* Must have a body mass index (BMI) of between 18 and 30 kg/m², inclusive
* Must have a body weight of not less than 50 kg
* Must have a blood pressure between 90 and 140 mmHg inclusive, systolic, and no higher than 90 mmHg diastolic at screening
* Must have normal renal function and no evidence of kidney damage (including abnormalities in blood or urine tests)

Exclusion Criteria:

* History of or current clinically significant medical illness
* Use of any systemic prescription or nonprescription medication (including vitamins and herbal supplements)
* Known allergy to canagliflozin or metformin or any of the excipients of the formulation
* Known allergy to heparin or history of heparin induced thrombocytopenia
* History of smoking or use of nicotine-containing substances within the previous 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of canagliflozin following the dose of 2 CANA/MET XR FDC tablets | Day 1, Day 7
  Plasma concentrations of canagliflozin are used to evaluate how long canagliflozin stays in the body.
Plasma concentration of metformin following the dose of 2 CANA/MET XR FDC tablets | Day 1, Day 7
  Plasma concentrations of metformin are used to evaluate how long it stays in the body.

SECONDARY OUTCOMES:
Percentage of participants with adverse events as a measure of safety and tolerability | Screening, up to Day 10 of the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States